CLINICAL TRIAL: NCT05535647
Title: Second Line Therapy With Regorafenib and HAIC Compared to FOLFOX for Advanced Intrahepatic Cholangiocarcinoma
Brief Title: Second Line Therapy for Advanced Intrahepatic Cholangiocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E20220698
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: Intrahepatic Cholangiocarcinoma; Regorafenib; HAIC; FOLFOX
MeSH Terms: conditions — Cholangiocarcinoma | interventions — regorafenib; Folfox protocol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regorafenib and HAIC (Experimental): Regorafenib HAIC with FOLFOX
  Interventions: Drug: Regorafenib and HAIC
- FOLFOX (Active Comparator): FOLFOX
  Interventions: Drug: FOLFOX

INTERVENTIONS:
Drug: Regorafenib and HAIC — Regorafenib: oral 80mg/day, D1-21, Q28d; HAIC with FOLFOX: hepatic artery infusion Oxa 85 mg/m2, CF 400 mg/m2, 5-Fu 400 mg/m2, 5-Fu 2400mg/m2 infusion 48h.
  Arms: Regorafenib and HAIC
Drug: FOLFOX — Oxa 85 mg/m2, CF 400 mg/m2, 5-Fu 400 mg/m2, 5-Fu 2400mg/m2 infusion 48h.
  Arms: FOLFOX

SUMMARY:
This is a prospective, Two-arm, comparative, randomized, controlled phase II trial, to explore the efficacy and safety of Regorafenib and HAIC vs. FOLFOX as Second Line Therapy for Advanced Intrahepatic Cholangiocarcinoma.

DETAILED DESCRIPTION:
Currently, complete surgical resection represents the only potentially curative treatment option for cholangiocarcinoma (CCA, including intrahepatic, hilar and distal CCA) and gallbladder carcinoma (GBCA). However,only less than 25% of patients are resectable at diagnosis and, even in this subset of patients, relapse rate is high.

Cisplatin and gemcitabine combination was identified as the standard first-line chemotherapy, yielding a median progression free survival (PFS) and median OS of 8.5 and 11.7 months, respectively. FOLFOX was the standard second-line chemotherapy. But the benefit of FOLFOX was limited.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated IRB/IEC-approved Informed Consent.
* Cytological or histological diagnosis of locally advanced or metastatic adenocarcinoma of the Intrahepatic Cholangiocarcinoma.
* Disease progressing after first-line chemotherapy with gemcitabine and platinum analogs (only one prior systemic therapy allowed).
* Age 18-75 years
* Karnofsky Performance Status > 50%
* Estimated life expectancy of at least 3 months.
* Negative pregnancy test (if female in reproductive years).
* Adequate bone marrow, liver and kidney function: leukocyte > 3500/mm3; absolute neutrophil count (ANC) > 1500/mm3; platelet count > 100000/mm3; hemoglobin > 10 g/dl; creatinine < 1.5 mg/dL; total bilirubin ≤ 1.5 x upper limit of normal range (ULN); SGOT e SGPT ≤ 2.5 ULN
* At the time of start of treatment, at least 2 weeks must have elapsed since completion of prior chemotherapy, minor surgery and radiotherapy (provided that no more than 25% of bone marrow reserve has been irradiated).
* Resolution of all acute toxic effects of any prior chemotherapy, surgery or radiotherapy to NCI CTC (Version 4.03) grade ≤ 1 for hematologic toxicities and ≤ 2 for non hematologic toxicities, with the exception of alopecia.
* Able and willing to comply with scheduled visits, therapy plans, and laboratory tests required in this protocol.

Exclusion Criteria:

* History of cardiac disease
* Ongoing infection > Grade 2 according to NCI-CTCAE version 4.03. Hepatitis B is allowed if no active replication (defined as abnormal ALT >2xULN associated with HBV DNA >20,000 IU/mL) is present
* Severe co-morbid illness and/or active infections including active hepatitis C and human immunodeficiency virus (HIV) infection
* History of interstitial lung disease (ILD).
* Any cancer curatively treated < 3 years prior to study entry, except cervical carcinoma in situ, treated basal cell carcinoma, and superficial bladder tumors (Staging: Ta, Tis and T1).
* Renal failure requiring hemo- or peritoneal dialysis.
* Clinically significant GI bleeding (CTCAE 4.03 grade 3 or higher) within 30 days prior to start of screening
* Thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks) within 6 months prior to start of screening.
* History of organ allograft, cornea transplantation will be allowed
* Active CNS metastases not controllable with radiotherapy or corticosteroids Visible retinal pathology as assessed by ophthalmologic exam that is considered a risk factor for RVO or CSR.
* Known history of hypersensitivity to study drugs
* Non-healing wound, ulcer, or bone fracture.
* Patients with seizure disorder requiring medication.
* Acute steroid therapy or taper for any purpose (chronic steroid therapy is acceptable provided that the dose is stable for 1 month before start of screening and thereafter).
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
* Pregnant or lactating women. Women of childbearing potential not employing adequate contraception. Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to start of study treatment and a negative result must be documented before first dose of study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-25 (Estimated); Primary Completion 2024-09-25 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 12month
  the rate of complete response and partial response among all evaluable patients

SECONDARY OUTCOMES:
Disease control rate (DCR) | 12 months
  the rate of complete response, partial response and stable disease among all evaluable patients
Progression-free Survival (PFS) | 12 months
  A duration from the date of initial treatment to disease progression (defined by RECIST 1.1) or death of any cause.
Overall Survival (OS) | 24 months
  Duration from the date of initial treatment to the date of death due to any cause.
Adverse events (AE) | 24 months
  Adverse events in each cycle were documented based on CTCAE v 4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No